CLINICAL TRIAL: NCT00784446
Title: A Phase I/II Study of Capecitabine/Oxaliplatin (XELOX) in Combination With Bevacizumab and Imatinib as First-line Treatment of Patients With Stage IV Colorectal Cancer
Brief Title: First-line Therapy of Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Roche Pharma AG (Industry); Novartis (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Ulrich Hacker, PD Dr., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO KRK 0205; ML20344
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Stage IV Colorectal Cancer
Keywords: AIO; colorectal cancer; 0205; Capecitabine; Oxaliplatin; Bevacizumab; Imatinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Bevacizumab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XELOX, Bevacizumab, Imatinib (No Intervention)
  Interventions: Drug: Oxaliplatin, Capecitabine, Bevacizumab, Imatinib

INTERVENTIONS:
Drug: Oxaliplatin, Capecitabine, Bevacizumab, Imatinib — Dose level I:
  Bevacizumab day 1: 7,5 mg/kg body weight Oxaliplatin day 1: 100 mg/m2 Capecitabine days 1-14 bid: 800 mg/m2 Imatinib days 1-21: 300 mg
  Repeat on day 22.
  Dose level II:
  Bevacizumab day 1: 7,5 mg/kg body weight Oxaliplatin day 1: 130 mg/m2 Capecitabine days 1-14 bid: 1000 mg/m2 Imatinib days 1-21: 300 mg
  Repeat on day 22.
  Other Names: Xeloda; Avastin; Imatinib; Eloxatin

SUMMARY:
Assessment of safety and toxicity, definition of the dose limiting toxicity (DLT) of the combination therapy consisting of Capecitabine, Oxaliplatin, Bevacizumab and Imatinib.

DETAILED DESCRIPTION:
The monoclonal anti-VEGF antibody bevacizumab has been approved for the treatment of stage IV colorectal cancer. The tyrosine kinase inhibitor imatinib mesylate has been shown to efficiently target PDGF-signalling. Blocking PDGFR-signalling leads to disruption of pericytes from the endothelium and reverses the maturation status thereby enhancing the sensitivity to anti-VEGF therapy.This background forms a rationale for a combined therapeutic PDGF and VEGF inhibition. Since bevacizumab shows best activity when used in combination with chemotherapy, capecitabine and oxaliplatin are included in this protocol. Patients with stage IV colorectal cancer and no prior chemotherapy can enter the study. Patients receive oral imatinib once a day on days 1-21. Oral Capecitabine is given on days 1-14 bid, Oxaliplatin and Bevacizumab are given on day 1. Courses are repeated every 22 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven inoperable colorectal cancer
* Adult patients >= 18 years of age
* ECOG <2

Exclusion Criteria:

* Preceding chemo- or immunotherapy with the exception of adjuvant or neoadjuvant treatment of non-metastatic disease ending ≥ 6 month prior to study inclusion. Progression within 6 month after the end of adjuvant therapy must be excluded.
* Other malignancies with the exception of basal cell carcinoma or successfully treated carcinoma in situ of the cervix uteri.
* No history of severe comorbidities, i. e. uncontrolled hypertension, GI-bleeding, congestive heart-failure NYHA class II-IV, symptomatic coronary heart disease, myocardial infarction within 1 year prior to study inclusion, serious cardiac arrhythmias requiring medication, Grade II or greater peripheral vascular disease and other severe uncontrolled co-morbidities
* No history of stroke or other CNS-diseases (tumors, seizure, transient ischemic attack etc.)
* ≥ Grade II peripheral artery vascular occlusive disease
* Preexisting neuropathy ≥ Grade 1
* Interstitial pneumonia or lung fibrosis
* Serious, nonhealing wound, ulcer, or bone fracture
* Preceding irradiation an indicator lesion except for documented progressive disease during irradiation and termination of irradiation ≥ 4 weeks from study inclusion
* Thromboembolic or bleeding events within the last 6 month
* Need for therapeutic anticoagulation (heparin, cumarin)
* Use of ASS > 325 mg/die or NSAR
* Proteinuria > 1+ (stix) as long as urine protein >1g/24h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity. | 6 weeks

SECONDARY OUTCOMES:
Assessment of overall response rate and progression free survival. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Hacker, PD Dr., Principal Investigator — University Cologne
Locations (8):
- Germany (8):
  - Medical Clinic for Haematology and Oncology, Cologne, North Rhine-Westphalia
  - Städische Kliniken Esslingen, Esslingen am Neckar
  - Klinikum St. Georg gGmbH, Leipzig
  - Johannes-Gutenberg-Universität Mainz, Mainz
  - Klinikum Mannheim, Mannheim
  - Prosper-Hospital, Recklinghausen
  - Leopoldina Krankenhaus, Schweinfurt
  - Universitätsklinik Ulm, Ulm